CLINICAL TRIAL: NCT00449553
Title: A Prospective Study of Associations of Changes in HbA1C and Fasting Blood Lipids Due to Treatment With Pioglitazone for 6 Months and Genetic Polymorphism's in PPAR-gamma
Brief Title: Observational Study to Assess Glycosylated Hemoglobin Changes After 6 Months of Treatment With Pioglitazone.
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: H6E-CP-GLAR; U1111-1114-2473 (Registry Identifier: WHO)
Record Dates: First submitted 2007-03-01; First posted 2007-03-20 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; Sulfonylurea Compounds; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA-analyses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pioglitazone 15 mg QD + Sulphonylurea
  Interventions: Drug: Pioglitazone and sulphonylurea
- Pioglitazone 30 mg QD + Sulphonylurea
  Interventions: Drug: Pioglitazone and sulphonylurea
- Pioglitazone 15 mg QD + Metformin
  Interventions: Drug: Pioglitazone and metformin
- Pioglitazone 30 mg QD + Metformin
  Interventions: Drug: Pioglitazone and metformin

INTERVENTIONS:
Drug: Pioglitazone and sulphonylurea — Pioglitazone 15 mg, tablets, orally, once daily and stable sulphonylurea therapy for up to 24 months.
  Other Names: ACTOS®; AD4833
  Groups: Pioglitazone 15 mg QD + Sulphonylurea
Drug: Pioglitazone and sulphonylurea — Pioglitazone 30 mg, tablets, orally, once daily and stable sulphonylurea therapy for up to 24 months.
  Other Names: ACTOS®; AD4833
  Groups: Pioglitazone 30 mg QD + Sulphonylurea
Drug: Pioglitazone and metformin — Pioglitazone 15 mg, tablets, orally, once daily and stable metformin therapy for up to 24 months.
  Other Names: ACTOS®; AD4833
  Groups: Pioglitazone 15 mg QD + Metformin
Drug: Pioglitazone and metformin — Pioglitazone 30 mg, tablets, orally, once daily and stable metformin therapy for up to 24 months.
  Other Names: ACTOS®; AD4833
  Groups: Pioglitazone 30 mg QD + Metformin

SUMMARY:
The purpose of this study is to asses changes in glycosylated hemoglobin, fasting blood lipids and genetic polymorphism's in peroxisomal proliferator activated receptors--gamma receptor after 6 months of pioglitazone, once daily (QD), treatment.

DETAILED DESCRIPTION:
The metabolic control in type 2 diabetes mellitus can be measured by means of glycosylated hemoglobin. A low value glycosylated hemoglobin indicates a good metabolic control, and has been shown to be associated with a better prognosis regarding diabetic complications. Type 2 diabetes is a disease with a profound genetic component. Peroxisome proliferator-activated receptor gamma is a transcription factor implicated in adipocyte differentiation, lipid and glucose metabolism. Peroxisome proliferator-activated receptor alfa is a transcription factor implicated in lipid oxidation and gluconeogenesis and is present in liver, kidney, heart, skeletal muscle and adipose tissue.

Pioglitazone is a thiazolidinedione that targets nuclear peroxisomal proliferator activated receptors, members of the super family of ligand activated transcription factors. Specifically, thiazolidinediones bind to the peroxisome proliferator-activated receptor gamma and affect transcription factors that influence expression of genes responsible for the production of proteins important in carbohydrate and lipoprotein metabolism. These include increases in glucose transporters 1 and 4 resulting in enhanced peripheral glucose utilization by fat and skeletal muscle.

This is a pharmacoepidemiological study to evaluate whether the individual genotype of the patients have any influence on the efficacy of pioglitazone.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills all requirements for treatment with pioglitazone.
* Willing to start treatment with pioglitazone.

Exclusion Criteria:

* Has previously participated in this study.
* Is currently taking or have taken oral antidiabetic medications other than sulfonylurea or metformin within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving pioglitazone therapy.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2001-06; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin. | 6 months

SECONDARY OUTCOMES:
Change from baseline in Clinical Laboratory Tests (alanine transaminase, hematocrit and hemoglobin). | End of Treatment
Change from baseline in Body Weight. | End of Treatment
Percentage of treatment responders defined as a patient with 0.6% decrease in HbA1C from baseline visit to final visit or accomplishment of a HbA1c value at or below 6.5%. | End of Treatment
Change from baseline in beta-cell function (Homeostasis model assessment). | End of Treatment
Change from baseline in insulin resistance (Homeostasis model assessment). | End of Treatment
Change from baseline in fasting lipoproteins (total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein-cholesterol and triglycerides). | End of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda Global Research and Developmnet Center Inc
Locations (4):
- Multiple, Denmark
- Multiple, Iceland
- Multiple, Norway
- Multiple, Sweden

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI